CLINICAL TRIAL: NCT01116544
Title: Treatment of Chronic Stroke With AMES + EMG Biofeedback
Acronym: AMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AMES Technology (Industry)
Collaborators: Oregon Health and Science University (Other); Emory University (Other); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT NS060192
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Stroke; Plegia; Paresis; Cerebrovascular Accident
Keywords: AMES device; Cerebrovascular Accident; Chronic Stroke; Rehabilitation; Upper Extremity; Biofeedback
MeSH Terms: conditions — Stroke; Paralysis; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMES therapy with EMG biofeedback (Experimental): The AMES device provides a 30 minute treatment period of alternating passive flexion and then extension of the hand while vibrators vibrate the muscles of the hand. The subjects job is to attempt to assist the device in the movement. A computer screen will provide visual feedback of the amount of EMG activity the subject is able to generate in the hand. This study will examine whether AMES therapy combined with EMG biofeedback can restore hand opening to plegic stroke subjects.
  Interventions: Device: AMES Therapy (assisted movement and enhanced sensation)
- AMES therapy with Torque biofeedback (Experimental): The AMES device provides a 30 minute treatment period of alternating passive flexion and then extension of the hand while vibrators vibrate the muscles of the hand. The subjects job is to attempt to assist the device in the movement. A computer screen will provide visual feedback of the amount of torque (force) the subject is able to generate in the hand during the movement. This study will examine whether AMES therapy combined with Torque biofeedback can restore hand opening to plegic stroke subjects.
  Interventions: Device: AMES Therapy (assisted movement and enhanced sensation)

INTERVENTIONS:
Device: AMES Therapy (assisted movement and enhanced sensation) — Each subject will receive 30 sessions of AMES therapy in the clinic. Each session will consist of 10 min of functional testing (i.e., passive motion and strength tests) followed by 30 min of grasp therapy using the AMES device. One group of subjects will receive AMES therapy only with joint torque biofeedback (without EMG feedback), and the other group will receive AMES therapy with EMG biofeedback. While all test subjects should attempt to open the hand when the grasp mechanism is opening and close the hand when the mechanism is closing, the biofeedback information provided to aid a subject will differ for the 2 subject groups.
  Other Names: Robotic

SUMMARY:
The purpose of this study is to determine if individuals who had a stroke more than one year before entering the study and who remain unable to open their affected hand are better able to sense and move their affected arm after 10-15 weeks of treatment with a new robotic therapy device (the AMES device) and EMG biofeedback.

DETAILED DESCRIPTION:
Over the last 20 years, the discovery of cortical plasticity in the adult human brain has led to the development of new therapies to rehabilitate stroke survivors whose recovery of motor function has stalled with conventional therapeutic methodology. However, the efficacy of these new therapies appears to be limited to relatively high-functioning chronic stroke patients. A therapeutic approach that may be efficacious in restoring functional movement to low-functioning chronic stroke patients is "AMES," which stands for Assisted Movement with Enhanced Sensation. Despite the efficacy of AMES in restoring movement to low-functioning hemiparetic stroke patients, those with plegia at a joint tend not to recover movement in the plegic direction with AMES treatment or with other rehabilitation therapies. The objective of this study is to determine if AMES treatment in combination with biofeedback can be helpful in restoring functional movement to plegic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Hemispheric stroke (ischemic or hemorrhagic), cortical or sub-cortical, documented by either a CT or MRI scan and associated with residual upper extremity weakness.
* Chronic stroke, occurring ≥12 months prior to subject enrollment.
* Age 18-80 years old.
* Inability to move any of the fingers of the affected hand more than 5.0 cm into extension.
* Finger-and-wrist impedance ≤3 on the Modified Ashworth Scale.
* Measureable EMG (>2 x baseline) in the long finger extensor muscle during attempted hand opening or closing.
* Physically and cognitively capable of consenting to and complying with the protocol (based on exam by Study Physician).
* Subject must be physically capable of communicating informed consent or must be accompanied by legally authorized representative to provide informed consent.

Exclusion Criteria:

* Complete flaccidity of the affected arm.
* Significant upper extremity proprioceptive deficit (<70% correct detection of the direction of passive finger movement with eyes closed).
* Pathological neurological/physical conditions, other than stroke, impairing the function of the impaired arm or resulting in pain in the arm.
* Spinal cord injury, arthritis, or fractures of affected arm that have resulted in loss of range of motion.
* Peripheral nerve injury or neuropathy resulting in significant motor or sensory loss in the tested arm.
* Cardiopulmonary compromise including but not limited to uncontrolled hypertension or angina, deep vein thrombosis, decompensated congestive heart failure, myocardial infarction, heart irregularities, or exercise intolerance.
* Major active psychiatric disorder.
* Cognitively or behaviorally unable to follow instructions including severe apraxia; inability to understand verbal (English) directions, or inability to communicate adequately with study personnel.
* Size of arm incompatible with the AMES device (checked by placing the limb in the device).
* Severe contractures or decreased range of motion or skin condition that would prohibit comfortable positioning or tolerance of the device or the vibrators.
* Any progressive neurodegenerative disorder affecting the upper extremity motor system.
* Uncontrolled seizure disorder.
* Current abuse of alcohol or drugs.
* Terminal illness with anticipated survival of <12 months.
* Current or planned concurrent participation in another study involving therapy to the impaired arm
* Planned initiation of or cessation of any kind of clinical therapy to the impaired limb just prior to or during the AMES treatment period.
* NIH Stroke Scale, following scores: Sensory Item score of >1; Neglect involving the affected limb score >1.
* Intent to receive Botox injections (5 months prior to or during enrollment), initiation of antispasmodic medication, or use of any other robotic (e.g., MANUS, Locomat) or electrical or vibratory stimulation device (e.g., Bioness) while participating in the AMES trial.
* Cognitively or behaviorally unable to follow instructions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-09-21 (Actual); Primary Completion 2011-02-28 (Actual); Study Completion 2011-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Cordo, PhD, Study Director — Oregon Health and Science University
Locations (3):
- United States (3):
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Oregon Health and Science University, Portland, Oregon

REFERENCES:
- [Derived] Cordo P, Wolf S, Lou JS, Bogey R, Stevenson M, Hayes J, Roth E. Treatment of severe hand impairment following stroke by combining assisted movement, muscle vibration, and biofeedback. J Neurol Phys Ther. 2013 Dec;37(4):194-203. doi: 10.1097/NPT.0000000000000023. PMID 24232364

RESULTS

PARTICIPANT FLOW:
Groups:
- AMES Therapy With EMG Biofeedback: The AMES device provides a 30 minute treatment period of alternating passive flexion and then extension of the hand while vibrators vibrate the muscles of the hand. The subjects job is to attempt to assist the device in the movement. A computer screen will provide visual feedback of the amount of EMG activity the subject is able to generate in the hand. Each subject will receive 30 sessions of AMES therapy in the clinic. Each session will consist of 10 min of functional testing (i.e., passive motion and strength tests) followed by 30 min of grasp therapy using the AMES device.
- AMES Therapy With Torque Biofeedback: The AMES device provides a 30 minute treatment period of alternating passive flexion and then extension of the hand while vibrators vibrate the muscles of the hand. The subjects job is to attempt to assist the device in the movement. A computer screen will provide visual feedback of the amount of joint torque the subject is able to generate in the hand. Each subject will receive 30 sessions of AMES therapy in the clinic. Each session will consist of 10 min of functional testing (i.e., passive motion and strength tests) followed by 30 min of grasp therapy using the AMES device.
Period: Overall Study
Arm/Group | AMES Therapy With EMG Biofeedback | AMES Therapy With Torque Biofeedback
Started | 23 | 23
Completed | 21 | 22
Not Completed | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Stroke ≥1 year post-injury with severe limitation of finger extension, but with intact upper limb proprioception.
Groups:
- Total: Total of all reporting groups
Arm/Group | AMES Therapy With EMG Biofeedback | AMES Therapy With Torque Biofeedback | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (13) | 45 (15) | 46 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 10 | 22
  White | 7 | 11 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Fugl-Meyer Assessment-Upper Limb [Mean (Standard Deviation); unit: units on a scale] — Measurement of impairment in the upper limb based on tone, range-of-motion, and synergies. Total score includes only the upper extremity portion of the Motor Function subscale of the assessment, that subset having a scoring range of 0-66, with 0 representing no function and no visible reflexes (i.e., profound plegia) and 66 representing normal motor function.
  units on a scale | 19.4 (6.2) | 23.1 (8.8) | 21.3 (7.8)
Strength Test Flexion [Median (Inter-Quartile Range); unit: Newton-meters] — Based on average strength in first 3 training sessions.
  Newton-meters | 16.6 [8.3 to 33.6] | 18.0 [13.4 to 31.6] | 17.6 [11.8 to 30.8]
Strength Test Extension [Median (Inter-Quartile Range); unit: Newton-meters] | -4.4 [-12.6 to -1.2] | 0.4 [-1.5 to 6.0] | -0.9 [-5.7 to 1.1]
Stroke Impact Scale (Physical Problems, Mobility, Hand, ADL) [Mean (Standard Deviation); unit: units on a scale] — Four of 8 possible subscales were used: Physical Problems, Mobility, Hand, and Daily Living, consisting of 26 total questions [scored from 1 (least impact) to 5 (most impact)]. The total (summed) raw score for all 4 sub-scales has a minimum of 26 and maximum of 130. The total raw score is then transformed:
  [(Actual Raw Score-Lowest Possible Raw Score)/Possible Raw Score Range] X 100. The minimum transformed score is 0 and the maximum is 100.
  units on a scale | 51.0 (9.1) | 53.6 (17.0) | 52.3 (9.1)
Stroke Impact Scale (Stroke Recovery) [Mean (Standard Deviation); unit: units on a scale] — A separate section of the Stroke Impact Scale measures self-perception of stroke recovery. Stroke recovery is based on a scale of 0-100, with 0 representing no recovery and 100 representing full recovery.
  units on a scale | 44.0 (23.3) | 48.0 (23.3) | 46.0 (23.1)
Box-and-Block Test [Median (Inter-Quartile Range); unit: Blocks moved] — Measure of functional movement
  Blocks moved | 0.0 [0.0 to 0.5] | 0.0 [0.0 to 2.75] | 0.0 [0.0 to 1.0]

OUTCOME MEASURES:

1. Primary Outcome: Box and Blocks Test
Description: Measurement of the change in functional movement of the hand associated with 30 AMES training sessions.
Time Frame: Within a week of completing all training sessions.
Population: Chronic stroke with severe hand impairment
Measure: Median (Inter-Quartile Range); unit: Number of blocks moved
Arm/Group | AMES Therapy With EMG Biofeedback | AMES Therapy With Torque Biofeedback
Number analyzed (Participants) | 21 | 22
Number of blocks moved | 0.0 [0.0 to 1.5] | 0.5 [0.0 to 5.25]
Statistical Analysis 1: Comparison: AMES Therapy With EMG Biofeedback vs AMES Therapy With Torque Biofeedback; Test type: Superiority or Other; p < 0.005, Wilcoxon (Mann-Whitney) — A priori threshold = 0.05

2. Secondary Outcome: Fugl-Meyer (UL) Assessment
Description: Scale: Fugl-Meyer Assessment-Motor Function-Upper Limb Measurement of impairment in the upper limb based on tone, range-of-motion, and synergies. Total score in this study includes only the Upper Limb portion of the Motor Function subscale of the assessment, the Upper Limb subset having a scoring range of 0-66, with 0 representing no function and no visible reflexes (i.e., profound plegia) and 66 representing normal motor function.
Time Frame: At baseline and again within a week of completing all training sessions. The interval between measurements was 10-12 weeks.
Population: Chronic stroke with severe upper limb impairment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMES Therapy With EMG Biofeedback | AMES Therapy With Torque Biofeedback
Number analyzed (Participants) | 21 | 22
units on a scale | 23.7 (6.2) | 27.0 (10.3)
Statistical Analysis 1: Comparison: AMES Therapy With EMG Biofeedback vs AMES Therapy With Torque Biofeedback; Test type: Non-Inferiority or Equivalence — Power analysis called for sample sizes of 32 participants in each treatment group. The study was close before reaching this number of participants; p < 0.001, ANCOVA — Hypothesis: significant increase in score (post-tx - pre-tx) for both groups; FMA scores adjusted for baseline differences

3. Secondary Outcome: Stroke Impact Scale (Physical Problems, Mobility, Hand, ADL)
Description: Four of 8 possible subscales were used: Physical Problems, Mobility, Hand, and Daily Living, consisting of 26 total questions [scored from 1 (least impact) to 5 (most impact)]. The total (summed) raw score for all 4 sub-scales has a minimum of 26 and maximum of 130. The total raw score is then transformed:
  [(Actual Raw Score-Lowest Possible Raw Score)/Possible Raw Score Range] X 100. The minimum transformed score is 0 and the maximum is 100.
Time Frame: Within a week of completing all training sessions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMES Therapy With EMG Biofeedback | AMES Therapy With Torque Biofeedback
Number analyzed (Participants) | 21 | 22
units on a scale | 54.0 (8.1) | 57.4 (18.0)
Statistical Analysis 1: Comparison: AMES Therapy With EMG Biofeedback vs AMES Therapy With Torque Biofeedback; Test type: Superiority or Other; p = 0.001, ANCOVA — Across both groups, whether score increased following completion of intervention

4. Secondary Outcome: Stroke Impact Scale (Stroke Recovery)
Description: A separate section of the Stroke Impact Scale measures self-perception of stroke recovery. Stroke recovery is based on a scale of 0-100, with 0 representing no recovery and 100 representing full recovery.
Time Frame: Within a week of completing all training sessions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMES Therapy With EMG Biofeedback | AMES Therapy With Torque Biofeedback
Number analyzed (Participants) | 21 | 22
units on a scale | 58.3 (18.2) | 63.3 (17.3)
Statistical Analysis 1: Comparison: AMES Therapy With EMG Biofeedback vs AMES Therapy With Torque Biofeedback; Test type: Superiority or Other; p = 0.001, ANCOVA — Across both treatment groups

5. Secondary Outcome: Strength Test Flexion
Description: Maximum squeezing (i.e., flexion) strength for thumb and fingers at the end of each training session. The participant squeezed the hand as hard as possible 3 times with a 5-10 second rest period between each effort. A single score was calculated for each training session as the average of the 3 efforts. Baseline score was based on the average of the first 3 session scores (i.e., 9 total efforts over the first 3 training sessions). Final score was based on the average of the last 3 training sessions.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Newton-meters
Arm/Group | AMES Therapy With EMG Biofeedback | AMES Therapy With Torque Biofeedback
Number analyzed (Participants) | 21 | 22
Newton-meters | 21.2 [10.4 to 30.9] | 30.8 [16.7 to 41.4]
Statistical Analysis 1: Comparison: AMES Therapy With EMG Biofeedback vs AMES Therapy With Torque Biofeedback; Data combined between 2 treatment groups; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Strength Test Extension
Description: Maximum opening (i.e., extension) strength for thumb and fingers at the end of each training session. The participant squeezed the hand as hard as possible 3 times with a 5-10 second rest period between each effort. A single score was calculated for each training session as the average of the 3 efforts. Baseline score was based on the average of the first 3 session scores (i.e., 9 total efforts over the first 3 training sessions). Final score was based on the average of the last 3 training sessions.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Newton-meters
Arm/Group | AMES Therapy With EMG Biofeedback | AMES Therapy With Torque Biofeedback
Number analyzed (Participants) | 21 | 22
Newton-meters | -11.4 [-17.7 to -0.8] | 0.6 [-0.2 to 2.8]
Statistical Analysis 1: Comparison: AMES Therapy With EMG Biofeedback vs AMES Therapy With Torque Biofeedback; Both treatment groups combined; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 2 years, 7 months
Description: Subjects were seen by the Trainer (i.e., treatment specialist) 2-3 times per week. At each training session, the Trainer routinely asked the subject whether he/she had experienced an event since the last session. If so, the occurrence and details were recorded in the Subject Progress Report for that training day. The Site Clinician subsequently made the determination of whether the serious or unanticipated events were related to the study procedures.
Arm/Group | AMES Therapy With EMG Biofeedback | AMES Therapy With Torque Biofeedback
Serious Adverse Events (participants affected / at risk) | 3/23 | 0/23
Other Adverse Events (participants affected / at risk) | 6/23 | 8/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMES Therapy With EMG Biofeedback (N=23) | AMES Therapy With Torque Biofeedback (N=23)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Fall not related to study
Scratched cornea (Eye disorders) | 1 (1) | 0 (0) — From contact lens, not related to study
Flu-like symptoms, high blood pressure (Cardiac disorders) | 1 (1) | 0 (0) — Treated at hospital, not related to study
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMES Therapy With EMG Biofeedback (N=23) | AMES Therapy With Torque Biofeedback (N=23)
Fall (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (2)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (2) — From vibrator
Muscle soreness/fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Hand pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No